CLINICAL TRIAL: NCT03642691
Title: A Treatment Protocol for Extended Administration of Prometic Plasminogen (Human) by Intravenous Infusion in Subjects With Hypoplasminogenemia Requiring Plasminogen Replacement Therapy
Brief Title: A Treatment Protocol for Expanded Access Administration of Prometic Plasminogen Due to Closure of Clinical Trial
Status: No longer available | Type: Expanded Access
Sponsor: Prometic Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2002C018G
Record Dates: First submitted 2018-08-10; First posted 2018-08-22 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Hypoplasminogenemia
MeSH Terms: conditions — Congenital Plasminogen Deficiency

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate, Treatment

INTERVENTIONS:
Biological: Ryplazim — Plasminogen IV replacement therapy

SUMMARY:
The clinical trial is no longer enrolling and is currently closing and Prometic will continue to provide Plasminogen (Human) under a treatment protocol to subjects in the United States (US) with hypoplasminogenemia requiring plasminogen replacement therapy who completed the End of Study visit in the following Prometic-sponsored clinical trials: 2002C011G, 2002C013G, 2002C016G, 2002C017G and 2002C019G.

DETAILED DESCRIPTION:
US adult and pediatric subjects with hypoplasminogenemia requiring plasminogen replacement therapy who completed the End of Study visit in the following Prometic-sponsored clinical studies: 2002C011G, 2002C013G, 2002C016G, 2002C017G and 2002C019G will continue to receive their repeat-dose study of Plasminogen (Human) under a treatment protocol. Approximately, 15 subjects will be enrolled in the treatment protocol under an expanded access to continue to receive Plasminogen (Human) at a dose of 6.6 mg/kg as a 10 to 30-minute intravenous (IV) infusion at site visits or at home by either the subject or caregiver at the same frequency as in their prior Prometic-sponsored clinical study. Subjects or caregivers may be trained for study drug administration as deemed appropriate by the Investigator. Dosing frequency will be adjusted by the Investigator based on clinical response and plasminogen activity trough levels.

Subjects who completed the End of Study visit in studies 2002C011G, 2002C013G, 2002C016G, 2002C017G and 2002C019G and signed informed consent (and assent, if applicable) for the present study will be enrolled in this study; this visit will be designated as Day 1 of the present study. Subjects will return to their study site every 26 weeks, or more often as determined by the Investigator, for safety assessments and measurements of plasminogen activity trough levels at the Investigator's discretion.

Treatment with Plasminogen (Human) will continue until the product has been approved and is commercially available or discontinued at any time by the Sponsor or at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the criteria below to participate in this study:

  1. The subject or the subject's caregiver has provided informed consent (as well as assent by subjects with ages dictated by local Investigational Review Board [IRB] guidelines).
  2. Subject has a diagnosis of hypoplasminogenemia requiring replacement therapy with Plasminogen (Human).
  3. Subject has completed the End of Study visit at a United States site in the following Prometic-sponsored clinical studies: 2002C011G, 2002C013G, 2002C016G, 2002C017G and 2002C019G.
  4. Female and male subject agrees to use contraceptive methods from Day 1 through 14 days after last dose of study treatment (unless documented as biologically or surgically sterile [e.g., postmenopausal, vasectomized]), or has not reached reproductive age.

Exclusion Criteria:

* Subjects who are pregnant and/or lactating are excluded from participating in the study.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Lorber, MD, Principal Investigator — Tower Hematology, Oncology; Heather McDaniel, MD, Principal Investigator — Vanderbilt Childrens Hospital
Locations (3):
- United States (3):
  - Tower Hematology and Oncology, Beverly Hills, California
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Vanderbilt University Medical Center, Nashville, Tennessee